CLINICAL TRIAL: NCT02630030
Title: Phase 0 Analysis of Ixazomib (MLN9708) in Patients With Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Jeffrey James Olson, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00083003; NCI-2015-01682 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16071 (Other: Takeda); Winship3017-15 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib (Experimental): Patients receive ixazomib PO 3 hours before surgery.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Given PO
  Other Names: MLN9708

SUMMARY:
This phase 0 trial studies ixazomib citrate in treating patients with glioblastoma that has spread or returned after period of improvement who are planning to undergo surgery. When given by mouth, ixazomib may be able to reach tumor cells in the brain. Studying samples of tissue, blood, and plasma in the laboratory from patients receiving ixazomib may help doctors learn more about the effects of ixazomib on the cells. It may also help doctors understand how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measurement of tissue concentration of ixazomib (ixazomib citrate) in a glioblastoma after preoperative administration.

II. Measurement of blood and plasma concentration of ixazomib during surgical sampling after preoperative administration.

SECONDARY OBJECTIVE:

I. Assessment of the safety of ixazomib after single dose administration in glioblastoma patients undergoing surgery for tissue concentration assessment.

OUTLINE:

Patients receive ixazomib orally (PO) 3 hours before surgery.

After completion of study, patients are followed up for 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Patients must have a previous diagnosis of a recurrent or progressive glioblastoma for which surgical resection is now indicated
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2 or (Karnofsky performance status of 60 or above)
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³; platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Hemoglobin > 9 g/dL
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN for the lab utilized
* Creatinine ≤ 1.5 mg/dL
* Calculated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (ie, ≤ grade 1 toxicity) from the reversible effects of prior chemotherapy
* Major surgery, including craniotomy, within 14 days before enrollment
* Radiotherapy of brain tumor within 3 months before enrollment
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of cytochrome P450, family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of ginkgo biloba or St. John's wort
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has ≥ grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Participation in other clinical trials utilizing other therapeutic investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Quillin J, Patel R, Herzberg E, Alton D, Bikzhanova G, Geisler L, Olson J. A phase 0 analysis of ixazomib in patients with glioblastoma. Mol Clin Oncol. 2020 Nov;13(5):43. doi: 10.3892/mco.2020.2114. Epub 2020 Aug 13. PMID 32874573
- See also: Molecular and Clinical Oncology Publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7453381/pdf/mco-13-05-02114.pdf.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixazomib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] — The measure of dispersion data are not available. All efforts were made to obtain these data from the PI and the study documentation.
  Years | 50.33 (NA) — There is no standard deviation for this trial
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Ixazomib in Tumor Tissue
Description: The relationship between patient's demographic, tumor and drug concentration results will be assessed with Pearson's correlation coefficient and tested with Wald's test. In addition, the mean and standard error of the concentrations will be estimated using a random-effects model to account for the within-patient correlation of the tumor biopsy samples. Given the limited number of observations, a relatively simple covariance matrix (e.g. compound symmetry) will be assumed.
Time Frame: At time of surgery, approximately 3 hours
Population: Each participant's sample was analyzed separately. For participant 3, 3 samples were collected and analyzed in order to account for intratumor variability
Measure: Number; unit: ng/g
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
ng/g
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 7.88
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.03
  Participant 3 Sample 1: number analyzed (Participants) | 1
  Participant 3 Sample 1 | 4.17
  Participant 3 Sample 2: number analyzed (Participants) | 1
  Participant 3 Sample 2 | 2.70
  Participant 3 Sample 3: number analyzed (Participants) | 1
  Participant 3 Sample 3 | 3.25

2. Primary Outcome: Concentration of Ixazomib in Tumor Tissue
Description: as for outcome 1
Time Frame: At time of surgery, approximately 3 hours
Population: Each participant's plasma concentration was analyzed separately.
Measure: Number; unit: ng/g
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
ng/g
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 21.8
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 18.0
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 36.2

3. Primary Outcome: Number of Patients With Safety and Tolerability of Ixazomib
Description: Safety was assessed with routine postoperative laboratory, vital sign, neurologic exam, and imaging studies through the day of surgery to staple or suture removal. This data was collected and any adverse events graded and their relationship to ixazomib administration determined.
Time Frame: At the time of surgery, approximately 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) was used to stratify any adverse patient response to ixazomib. There were no clinically relevant adverse events as a result of ixazomib administration.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events collected through study completion, 30 days after study drug administration.
Arm/Group | Ixazomib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=3)
Anemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Immune system disorders) | 1
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Lipase (General disorders) | 1
Confusion (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT02630030/Prot_SAP_000.pdf